CLINICAL TRIAL: NCT06356012
Title: Immunophenotyping, Microbiome, Clinical Outcome and Biomarkers for Predicting Immunological Response in Patients with High-grade Cervical Intraepithelial Lesions Treated with Imiquimod
Brief Title: Clinical Outcome and Biomarkers for Predicting Immunological Response in Patients Treated with Imiquimod
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Farmoquimica S.A. (Industry); Hospital de Cancer de Barretos - Fundacao Pio XII (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 71163523.1.0000.5437
Record Dates: First submitted 2024-03-04; First posted 2024-04-10 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-04

CONDITIONS: HSIL, High-Grade Squamous Intraepithelial Lesions; Vaginal Microbiome; Biomarkers
MeSH Terms: conditions — Squamous Intraepithelial Lesions | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Imiquimod treatment plus Loop Electrosurgical Excision Procedure (Experimental): 36 patients diagnosed with CIN 3 who will be undergone 16 applications of 5g imiquimod twice a week and then Loop Electrosurgical Excision Procedure will procedure (60 days). Pathological analysis will evaluate the lesion histologically after immunomodulatory treatment. The individual's immunological response will also be evaluated during applications and after surgical intervention.
  Interventions: Drug: Imiquimod; Procedure: Loop Electrosurgical Excision Procedure
- Loop Electrosurgical Excision Procedure (Active Comparator): 30 patients diagnosed with CIN 3 who will be undergone Loop Electrosurgical Excision Procedure (60 days). Pathological analysis will evaluate the lesion histologically after treatment (LEEP). The individual's immunological response will also be evaluated after surgical intervention.
  Interventions: Procedure: Loop Electrosurgical Excision Procedure
- healthy population (No Intervention): Immunological markers will be evaluated in a healthy population that had negative screening tests for cervical lesions to compare to the population in the injury and intervention groups.

INTERVENTIONS:
Drug: Imiquimod — Experimental group will be treated with 16 applications of imiquimod and subsequently LEEP.
  Other Names: IXIUM
  Arms: Imiquimod treatment plus Loop Electrosurgical Excision Procedure
Procedure: Loop Electrosurgical Excision Procedure — Active comparator group will be treated with LEEP.
  Other Names: LEEP
  Arms: Imiquimod treatment plus Loop Electrosurgical Excision Procedure; Loop Electrosurgical Excision Procedure

SUMMARY:
The goal of this clinical trial is to identify the immunophenotypic profile of the local immune response, the cervicovaginal microenvironment and the microbiological profile of women with CIN 3 treated with imiquimod. Participants will be divided in 3 groups: CIN 3 who will use 16 doses of imiquimod in the uterine cervix, applied twice a week and will be treated with LEEP procedure; 2) patients with CIN 3 who will undergo standard treatment with LEEP procedure; 3) patients with negative cytology and HPV (human papillomavirus) test. Blood and cervicovaginal lavage collections will be performed at different times, for comparisons between cellular response profiles to imiquimod during treatment and baseline levels in healthy patients.

DETAILED DESCRIPTION:
INTRODUCTION: High-grade intraepithelial lesions (CIN 2/3) are considered precursor lesions of cervical cancer, and its treatment involves destructive or excisional methods. Some studies have proven the efficacy of the immunomodulator imiquimod as a topical treatment for CIN 2/3 lesions. Imiquimod activates the innate immune response through dendritic cells, monocytes and macrophages, in addition to modulating the response pattern of T lymphocytes. Thus, the characterization of the immune response in the treatment with imiquimod in lesions caused by oncogenic HPV, may benefit women in a way that it is possible to measure the response of each patient, improving the understanding of its mechanism of action, directly impacting the efficacy and adverse events. caused by the drug. OBJECTIVES: To identify the immunophenotypic profile of the local immune response, the cervicovaginal microenvironment and the microbiological profile of women with CIN 3 treated with imiquimod. MATERIALS AND METHODS: It will be included 90 patients, 60 with high-risk HPV, diagnosed with CIN 3 and 30 patients with negative cytology and HPV. Patients will be divided into 3 groups: 1) patients with CIN 3 who will use 16 doses of imiquimod in the uterine cervix, applied twice a week; 2) patients with CIN 3 who will undergo standard treatment with Transformation Zone Excision (EZT); 3) patients with negative cytology and HPV. Blood and cervicovaginal lavage will be collected for immunophenotypic analysis (flow cytometry), quantification of immunological mediators (Cytometric Bead Array) and evaluation of the microbiome (MiniION). The results obtained will be correlated with the clinical and pathological data of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 25 and 45 years of age (reproductive age);
* High-risk HPV carriers;
* Residents less than 300 km from the city of Barretos-São Paulo;
* With a histological diagnosis of high-grade cervical squamous intraepithelial lesion (CIN 3), obtained through colposcopy-guided biopsy performed at the Barretos Cancer Hospital (HCB);
* Acceptance of the Informed Consent Form.

Exclusion Criteria:

* Suspicion of invasive squamous cell carcinoma or Adenocarcinoma (in situ or invasive) by colposcopy and/or cytology;
* Pregnant or breastfeeding;
* Immunodeficiency condition;
* Previous treatment for high-grade cervical squamous intraepithelial lesion;
* Who have been immunized for HPV;
* Have used antibiotics in the last 30 days

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with histological regression of High-grade squamous intraepithelial lesion (HSIL) | 3 years
  A satisfactory immunological response is expected after the application of the immunomodulator imiquimod twice a week for 8 weeks in patients with CIN 3, with the objective of histological regression of the high squamous intraepithelial lesion (HSIL), which will be confirmed histologically after performing the gold standard LEEP treatment, which will be made available to all patients with CIN 3 included in the study

SECONDARY OUTCOMES:
Correlation between vaginal microbiome and immunological response | 3 years
  Analysis of the vaginal microbiota and its correlation with the immunological response to imiquimod in CIN 3 lesions

CONTACTS AND LOCATIONS:
Locations (1):
- Barretos Cancer Hospital, Barretos, Brazil